CLINICAL TRIAL: NCT06620939
Title: The Effect of Levonorgestrel Intrauterine System in Preventing Endometrial Polyps Recurrence After Hysteroscopic Polypectomy: Protocol of a Multi-center Randomised Controlled Trial
Brief Title: The Effect of Levonorgestrel Intrauterine System in Preventing Endometrial Polyps Recurrence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Jian (Other)
Collaborators: Nanjing Maternity and Child Health Care Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai First Maternal and Infant Health Hospital affiliated to Tongji University Medical School (Other); RenJi Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhang Jian, Principal Investigator, International Peace Maternity and Child Health Hospital
Organization: International Peace Maternity and Child Health Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IIT-2024-19
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-08

CONDITIONS: Endometrial Polyp
Keywords: Endometrial polyp; Levonorgestrel intrauterine system

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LNG-IUS group (Experimental): Participants will receive Mirena placement after hysteroscopic polypectomy
  Interventions: Drug: Levonorgestrel Intrauterine System (LNG-IUS)
- Control group (No Intervention): Participants will receive none additional treatment after hysteroscopic polypectomy.

INTERVENTIONS:
Drug: Levonorgestrel Intrauterine System (LNG-IUS) — Participants in the intervention group will receive Mirena placement after hysteroscopic polypectomy
  Arms: LNG-IUS group

SUMMARY:
The goal of this clinical trial is to determine whether the LNG-IUS is more effective to that of expectant in preventing endometrial polyp recurrence after hysteroscopic polypectomy.

Researchers will compare LNG-IUS to expectant management to see if LNG-IUS works to reduce the recurrence rate of endometrial polyps.

Participants will:

Receive Mirena placement or not after hysteroscopic polypectomy； Be scheduled for a follow-up with TVCD to screen for endometrial polyps recurrence every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. （1）Women age 20 to 48 years old;
2. （2）Previous history of endometrial polypectomy;
3. （3）Postoperative pathology confirmed endometrial polyps；
4. （4）Women without fertility desire within 2 years；
5. （5）Signed informed consent.

Exclusion Criteria:

1. （1）Contraindications for a hysteroscopic polypectomy or LNG-IUS or not willing to receive this type surgery；
2. （2）Women who have a positive pregnancy test；
3. （3）A I and II type submucosal uterine leiomyoma, congenital uterine malformation, atypical endometrial polyps, a (suspected) malignancy, atypical endometrial cells, reproductive tract infections；
4. （4）Postoperative pathology confirmed non-endometrial polyps；
5. （5）Postoperative pathology confirmed endometrial proliferative diseases which need hormone drug therapy after surgery；
6. （6）Treatment with hormonal three months before surgery；
7. （7）The uterine cavity is more than 10 cm deep；
8. （8）Women with severe diseases；
9. （9）Women who were enrolled in another clinical study that could potentially impact the objectives of this study prior to their initial visit were excluded.
10. （10）Unable to cooperate with the study procedures for various reasons, such as language comprehension difficulties, mental illness, inability to travel to the study center, or poor compliance.

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 558 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Endometrial polyps recurrence rate | 2 years

SECONDARY OUTCOMES:
Side effects and complications | 2 years
Visual Analogue Scale (VAS) score for chronic pelvic pain | 2 years
  The minimum value of this scoring table is 0, and the maximum value is 10. The higher the score, the higher the degree of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — International Peace Maternity and Child Health Hospital

IPD SHARING:
Plan to Share IPD: No